CLINICAL TRIAL: NCT05762939
Title: Effectiveness of a Therapy Chatbot on Anxiety and Depressive Symptoms in Subclinical Young Adults: A Randomized Controlled Trial
Brief Title: Chatbot Intervention for Anxiety and Depressive Symptoms in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RID_FIDO_RCT_1
Record Dates: First submitted 2023-02-10; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; quality of life; loneliness
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot (Experimental): Intervention using a pre-release version of Fido (https://fido.aid.pl), Polish AI-based therapy chatbot.
  Interventions: Behavioral: Chatbot
- Control (book) (Active Comparator): Intervention using self-help materials - chapters from a popular book on cognitive therapy, including worksheets.
  Interventions: Behavioral: Control (book)

INTERVENTIONS:
Behavioral: Chatbot — Participants in this condition were asked to use Fido, a Polish therapy chatbot, for two weeks. No minimal requirements of usage time were enforced, but participants had to fill in five engagement check surveys during the intervention period. Each survey had to be completed in less than 24 hours.
  Arms: Chatbot
Behavioral: Control (book) — Participants in this condition were told to read selected chapters from a self-help book during the two-week intervention period. No minimal requirements of usage time were enforced, but participants had to fill in five engagement check surveys during the intervention period. Each survey had to be completed in less than 24 hours.
  Arms: Control (book)

SUMMARY:
This clinical trial compares the effects of using an artificial intelligence based therapy chatbot and a self-help book to lower anxiety and depressive symptoms. The therapy chatbot (named Fido) is an application delivering support for mental health via a conversation-like interface in a highly inflected language (Polish).

The team will recruit young people (aged 18-35) who currently struggle with anxiety and/or depression. The participants will use the chatbot or self-help materials for two weeks. Then, the researchers will check if using the chatbot or the book improved several aspects of mental health and the quality of life. Moreover, they will compare the groups for any differences in outcomes.

DETAILED DESCRIPTION:
The primary objective of this randomized controlled trial is to evaluate the effectiveness of a chatbot-delivered cognitive-behavioural intervention on anxiety and depressive symptoms (and their correlates, such as quality of life or feelings of loneliness) in a subclinical sample of about 80 participants.

The intervention results are compared to an active control intervention with popular self-help materials. Secondary objectives include the assessment and analysis of the human-chatbot therapeutic bond and general user experience.

The study uses a 2 x 3 mixed factorial design with two intervention arms (Fido chatbot vs self-help book) and three time points (T1: just prior to the intervention, T2: immediately after the intervention, T3: at a follow-up one month after the previous measurement). The primary intervention lasts two weeks.

All primary and secondary outcomes are assessed using self-administered online questionnaires in Polish. Each primary outcome measure is analyzed using a 2 (arms) x 2 (time points) ANOVA models with T1-T2 comparisons to test for the intervention effect and T1-T3 comparisons to check the stability of the intervention effect. Additional analyzes utilize standard NHST calculations and procedures (such as t-tests and correlation coefficients) alongside the conventional ⍺=.05 level.

Similarly to the previous research in this area, no blinding is used. Participants are informed about different conditions, but the research hypotheses are masked.

ELIGIBILITY:
Inclusion Criteria:

* declaring at least mild depressive or anxiety symptoms by achieving a total score of at least 16 points on Center for Epidemiologic Studies Depression Scale Revised or at least 50 points on Penn State Worry Questionnaire
* being able to visit the study site in Poznań (Poland) to complete all measurements

Exclusion Criteria:

* undergoing psychotherapy, coaching or psychopharmacological treatment
* being diagnosed with a neurological disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
CESD-R Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum score of the Polish version of the Center for Epidemiologic Studies Depression Scale Revised.
PHQ-9 Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum score of the Polish version of the Patient Health Questionnaire-9.
PSWQ Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum score of the Polish version of the Penn State Worry Questionnaire.
SWLS Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum score of the Polish version of the Satisfaction With Life Scale.
PANAS Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum scores of the Polish version of the Positive and Negative Affect Scale in two subscales (Positive and Negative Affect, separately).
STAI Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum score of the Polish version of the State-Trait Anxiety Inventory.
R-UCLA Score Change | Time point 1: Just prior to the intervention. Time point 2: Immediately after two weeks of the intervention. Time point 3: One month after the previous measurement (time point 2).
  The total sum score of the Polish version of the Revised UCLA Loneliness Scale.

OTHER OUTCOMES:
ACC Score | Time point 2: Immediately after two weeks of the intervention.
  The total sum score of the Polish version of the Acceptability E-scale. Used exclusively in the chatbot arm.
HCI Scores | Time point 2: Immediately after two weeks of the intervention.
  The total sum scores of six subscales from the Human-Computer Interaction Scale. Used exclusively in the chatbot arm.
LP Score | Time point 2: Immediately after two weeks of the intervention.
  Individual item scores from Language Pragmaticality Scale. Used exclusively in the chatbot arm.
WAI-SR Score | Time point 2: Immediately after two weeks of the intervention.
  The total sum score of the Polish version of the Working Alliance Inventory Short Revised. The Polish translation of this measure was developed by the research team. Used exclusively in the chatbot arm.
Psychoeducation Test Score | Time point 2: Immediately after two weeks of the intervention.
  The total sum score of the 12-item test which assessed the participants' acquired knowledge of psychoeducation topics.

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Michałowski, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities, Warsaw, Poland
Locations (1):
- Laboratory of Affective Neuroscience in Poznań, SWPS University of Social Sciences and Humanities, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data from all enrolled participants will be publicly available in the project's OSF repository.
Supporting Information: ICF, Analytic Code
Time Frame: IPD and supporting documents will be available as soon as research results are published.
Access Criteria: IPD and supporting documents will be publicly available.

REFERENCES:
- [Background] Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8. doi: 10.1016/j.apnr.2009.04.003. Epub 2009 Sep 18. PMID 20974066
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. Clin Psychol Psychother. 2010 May-Jun;17(3):231-9. doi: 10.1002/cpp.658. PMID 20013760
- [Background] Moshe I, Terhorst Y, Philippi P, Domhardt M, Cuijpers P, Cristea I, Pulkki-Raback L, Baumeister H, Sander LB. Digital interventions for the treatment of depression: A meta-analytic review. Psychol Bull. 2021 Aug;147(8):749-786. doi: 10.1037/bul0000334. PMID 34898233
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Koziara K. Assessment of depressiveness in population. Psychometric evaluation of the Polish version of the CESD-R. Psychiatr Pol. 2016 Dec 23;50(6):1109-1117. doi: 10.12740/PP/61614. English, Polish. PMID 28211550
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Kusier AO, Folker AP. The Satisfaction with Life Scale: Philosophical Foundation and Practical Limitations. Health Care Anal. 2021 Mar;29(1):21-38. doi: 10.1007/s10728-020-00420-y. Epub 2021 Jan 2. PMID 33386535
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Derived] Karkosz S, Szymanski R, Sanna K, Michalowski J. Effectiveness of a Web-based and Mobile Therapy Chatbot on Anxiety and Depressive Symptoms in Subclinical Young Adults: Randomized Controlled Trial. JMIR Form Res. 2024 Mar 20;8:e47960. doi: 10.2196/47960. PMID 38506892
- See also: OSF Preregistration — https://doi.org/10.17605/OSF.IO/2CQT3